CLINICAL TRIAL: NCT03691740
Title: Nightly Suppression of Contractions in At-Risk Pregnancies by the Infusion of Defused Blue Light
Brief Title: Uterine Contractions Under Blue Light
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: Kyndermed (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00031969
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Preterm Contractions
Keywords: circadian, melatonin, preterm labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Study group assignments will be placed in an opaque envelope which will be kept in the designated research area on Labor and Delivery. After informed consent is obtained, the coordinator will take one of the envelopes to determine the study group. The coordinator will not communicate with the care provide or the investigator regarding study group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Ocular light will be applied via a mask. The participants allocated to the experimental group will receive blue light
  Interventions: Device: Ocular light
- Control (Placebo Comparator): Ocular light will be applied via a mask. The participants allocated to the control group will receive red light
  Interventions: Device: Ocular light

INTERVENTIONS:
Device: Ocular light — A light mask to which small light emitting diode(LED) lights emitting a blue or red color light will be used to deliver ocular light

SUMMARY:
The objective in the current study is to test the hypothesis that nocturnal uterine contractions in preterm women can be suppressed by brief ocular exposure to blue light.The Olcese lab at Florida State University identified a novel interaction between the myometrial melatonin receptors and OT receptors in human myometrial cells (Sharkey et al. 2009), which may ultimately help to resolve certain issues surrounding idiopathic preterm labor. Their results consistently indicate that melatonin at physiological concentration sensitizes human myometrial smooth muscle cells to the contractile effects of OT (Sharkey et al. 2010).

DETAILED DESCRIPTION:
Study participants will be pregnant women (gestational weeks 24 to 31+6 days) who present with preterm contractions. In the triage room, the study participant will be connected to the external tocometer from at least 19:00h (7 PM) to the following morning at 07:00h. Room lighting will be kept dim.

Participants meeting inclusion criteria will be randomly allocated to blue light or red light. Baseline contractions will be measured. The allocated light mask will be applied for 2 intervals of 60 minutes each.There will be a 60 minute rest period after every 60 minute intervention period for comparison.

Other than the application of the light mask, all routine standards of care deemed warranted by the obstetric provider for proper treatment of preterm labor will be followed. (ie antenatal steroids, tocolytics).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Gestational age: 24 to 31 (+6 days) week of pregnancy
* Uterine contractions
* First episode of preterm labor

Exclusion Criteria:

* Visual impairment (legally blind)
* Multiple pregnancy
* Current progesterone treatment
* Preeclampsia
* Renal disease
* Current chlamydia or gonorrhea infections
* Cocaine or opiate use
* Nightshift work in the past week

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-06 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of contractions per hour | Immediately upon completion of intervention
  Number of contractions per hour

SECONDARY OUTCOMES:
Binary proportion of 4 or less compared to 5+ contractions per hour | Immediately upon completion of intervention
  Compare proportion proportions among each treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Judette M Louis, MD, Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

REFERENCES:
- [Background] Sharkey JT, Puttaramu R, Word RA, Olcese J. Melatonin synergizes with oxytocin to enhance contractility of human myometrial smooth muscle cells. J Clin Endocrinol Metab. 2009 Feb;94(2):421-7. doi: 10.1210/jc.2008-1723. Epub 2008 Nov 11. PMID 19001515
- [Background] Olcese J, Beesley S. Clinical significance of melatonin receptors in the human myometrium. Fertil Steril. 2014 Aug;102(2):329-35. doi: 10.1016/j.fertnstert.2014.06.020. Epub 2014 Jul 9. PMID 25015556
- [Background] Olcese J, Lozier S, Paradise C. Melatonin and the circadian timing of human parturition. Reprod Sci. 2013 Feb;20(2):168-74. doi: 10.1177/1933719112442244. Epub 2012 May 3. PMID 22556015
- [Background] Sharkey JT, Cable C, Olcese J. Melatonin sensitizes human myometrial cells to oxytocin in a protein kinase C alpha/extracellular-signal regulated kinase-dependent manner. J Clin Endocrinol Metab. 2010 Jun;95(6):2902-8. doi: 10.1210/jc.2009-2137. Epub 2010 Apr 9. PMID 20382690